CLINICAL TRIAL: NCT01301859
Title: Treatment Initiation and Participation Program (TIP)
Brief Title: Personalized Antidepressant Adherence Strategies For Depressed Elders
Acronym: TIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Michigan (Other)
Responsible Party: Principal Investigator, Jo Anne Sirey, Associate Professor, Weill Medical College of Cornell University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01MH087562-01A1 (NIH); 1R01MH087562-01A1 (NIH)
Record Dates: First submitted 2011-02-18; First posted 2011-02-23 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Depression
Keywords: older adults; adherence; antidepressant; depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TIP Adherence Intervention (Active Comparator): The TIP program is a brief, individualized intervention designed as an adjunct to pharmacotherapy for depression prescribed by a primary care physician. The key to the intervention is the involvement of the older adult in creating an adherence strategy tailored to his/her barriers and needs.
  Interventions: Behavioral: TIP
- Usual Care (Placebo Comparator): Treatment as usual in a primary care setting
  Interventions: Behavioral: TIP

INTERVENTIONS:
Behavioral: TIP — Treatment visits as usual with MD

SUMMARY:
The study is a randomized controlled trial to test the usefulness of a brief intervention to improve adherence to antidepressant medication prescribed to older adults in a primary care setting. Study will be conducted at Weill Cornell and University of Michigan.

DETAILED DESCRIPTION:
The intervention is a brief, psychosocial intervention designed to be an adjunct to pharmacotherapy prescribed by a primary care physician. It includes psychoeducation, problem solving and development of goals and a personalized adherence strategy. The intervention includes three 30 minute sessions during the first 6 weeks of treatment and a follow-up phone call two weeks later.

ELIGIBILITY:
Inclusion Criteria:

Age: 65 and older; Newly prescribed antidepressant medication by PCP (within past 10 days); Has not been prescribed antidepressant medication in previous 6 months.

Exclusion Criteria:

High suicide risk, i.e. intent or plan to attempt suicide Presence of alcohol abuse, substance abuse, psychotic disorder or, bipolar disorder as observed on the SCID, are excluded; Dementia: MMSE below 24, clinical assessment, or medication; Inability to speak English; Aphasia interfering with communication; Terminal illness or current chemotherapy

-

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 231 (Actual)
Dates: Start 2011-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Brief Medication Questionnaire | 12 week Follow up
  Participants randomized to the TIP intervention will be significantly more likely to be adherent (take more than 80% of prescribed doses) to antidepressant treatment at 6-week follow-up (immediately after the intervention is completed) and 12-week follow-up (6 weeks after intervention is completed) as compared to older adults randomized to the Treatment as usual control condition.

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale | 12 weeks
  Participants randomized to the TIP intervention will have a significantly greater reduction of depressive symptoms (on the HDRS) from baseline to the 6-week, 12-week and 24-week follow-ups than older adults who are randomized to the treatment as usual control condition.

CONTACTS AND LOCATIONS:
Overall Officials: JoAnne Sirey, Ph.D., Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- United States (2):
  - University of Michigan, Ann Arbor, Michigan
  - Weil Cornell Medical College, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sirey JA, Banerjee S, Marino P, Bruce ML, Halkett A, Turnwald M, Chiang C, Liles B, Artis A, Blow F, Kales HC. Adherence to Depression Treatment in Primary Care: A Randomized Clinical Trial. JAMA Psychiatry. 2017 Nov 1;74(11):1129-1135. doi: 10.1001/jamapsychiatry.2017.3047. PMID 28973066